CLINICAL TRIAL: NCT04184687
Title: Randomized Study on the Treatment of Cartilaginous Lesions and Concomitant Anterior Cruciate Ligament Reconstruction
Brief Title: The Treatment of Cartilaginous Lesions and Concomitant Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CART-LCA
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cruciate Ligament Rupture; Cartilage Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanofractures treatment of the cartilaginous lesions (Experimental): Patients undergoing to anterior cruciate ligament reconstruction with concomitant treatment of the cartilaginous lesions with nanofractures technique.
  Interventions: Procedure: Nanofractures
- no treatment of the cartilaginous lesions (Active Comparator): Patients undergoing to anterior cruciate ligament reconstruction. Cartilaginous lesions won't be treated
  Interventions: Procedure: no treatment cartilaginous lesions

INTERVENTIONS:
Procedure: Nanofractures — anterior cruciate ligament reconstruction will be performed in combination with the nanofractures for the treatment of cartilaginous lesions
  Arms: Nanofractures treatment of the cartilaginous lesions
Procedure: no treatment cartilaginous lesions — patient undergoing to the anterior cruciate ligament reconstruction without treatment of the cartilaginous lesions
  Arms: no treatment of the cartilaginous lesions

SUMMARY:
The aim of the study is the evaluation of both clinical and radiological results in patients undergone to cruciate ligament reconstruction with concomitant cartilaginous lesion treated with or without nanofractures.

DETAILED DESCRIPTION:
The anterior cruciate ligament lesion is one of the most common disease conditions in the orthopedic clinical practice. The mechanism of injury is due to a direct or indirect knee trauma causing both ligamentous breaking and surface articular stress, with cartilaginous lesion often associated to the lesion of the anterior cruciate ligament.

The treatment of these lesions in combination with the treatment of the anterior cruciate ligament is controversial, more controversial is to understand the indication to treatment for these lesions.

In order to clarify this aspect and provide a more reliable therapeutic indication for the treatment of the cartilaginous lesion with concomitant anterior cruciate ligament lesion we want to compare the clinical outcomes of the non-treated cartilaginous lesions against the treated cartilaginous lesions wiht nonofractures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 18 < age < 55;
2. Patients with complete ACL injury candidates for surgical reconstruction of the same;
3. Cartilaginous lesion of the femur-tibial compartment of grade III-IV ICRS ≤3 cm2 confirmed intra-operatively;
4. Patients without evidence of osteoarthritis
5. Patients' ability and consent to participate in clinical and radiological follow-up;
6. Signature of informed consent.

Exclusion Criteria:

1. Patients incapable of understanding and of wanting;
2. State of immunodepression;
3. Patients with malignant neoplasms;
4. Patients suffering from rheumatic diseases;
5. Patients suffering from non-compensated diabetes;
6. Patients suffering from uncompensated thyroid metabolic disorders;
7. Patients abusing alcoholic beverages, drugs or drugs;
8. Patients with axial deviations> 5 °;
9. Body Mass Index> 35;
10. Patients treated with surgery at the same knee in the previous 12 months.
11. Cartilaginous lesions grade I-II according to the ICRS score.
12. Cartilage lesions with a diameter greater than 3 cm².
13. Non-suturable meniscal lesions requiring meniscectomy> 50% and patients with previous meniscectomies> 50% in the same compartment.
14. Need for further associated surgical procedures in addition to the reconstruction of ACL and possibly the nanofractures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2027-07-25 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
IKDC-subjective score (International Knee Documentation Committee) | 24 month
  It is a specific subjective rating scale for te knee. Iti s one of the most reliable tools for assessing knee diseases. The survey examines three categories: symptoms, sport activity, knee function.
WORMS (Whole-Organ Magnetic Resonance Imaging Score) | 24 month
  Magnetic resonance imaging will be evaluated through WORMS. The score evaluated five aspects of the three knee compartments (cartilage, bone marrow abnormalities, bone cysts, bone attrition and osteophytes) as well as the soft tissue (menisci, ligaments and synovium)

SECONDARY OUTCOMES:
IKDC-subjective score (International Knee Documentation Committee) | 6, 12, 36 and 60 months
  It is a specific subjective rating scale for te knee. Iti s one of the most reliable tools for assessing knee diseases. The survey examines three categories: symptoms, sport activity, knee function.
Tegner Activity Level Scale | 6, 12, 24, 36 and 60 months
  Survey useful for assessing sport activity of the patient.
KOOS (Knee injury and Osteoarthritis Outcome Score ) | 6, 12, 24, 36 and 60 months
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale
EQ-5D (EuroQoL) Current Health Assessment | 6, 12, 24, 36 and 60 months
  It is a reliable tools for assessing quality of life of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Filardo G, de Caro F, Andriolo L, Kon E, Zaffagnini S, Marcacci M. Do cartilage lesions affect the clinical outcome of anterior cruciate ligament reconstruction? A systematic review. Knee Surg Sports Traumatol Arthrosc. 2017 Oct;25(10):3061-3075. doi: 10.1007/s00167-016-4097-y. Epub 2016 Apr 4. PMID 27043346
- [Background] Brophy RH, Zeltser D, Wright RW, Flanigan D. Anterior cruciate ligament reconstruction and concomitant articular cartilage injury: incidence and treatment. Arthroscopy. 2010 Jan;26(1):112-20. doi: 10.1016/j.arthro.2009.09.002. PMID 20117635